CLINICAL TRIAL: NCT05160246
Title: Investigation of the Instant Effect of Kinesiology Taping on Rectus Femoris Muscle on Muscle Activation, Physical Performance and Proprioception in Knee Osteoarthritis Patients
Brief Title: The Instant Effect of Kinesiology Taping in Patients With Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Aylin Ataş, Principal investigator, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kinesiotape in Knee OA
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis, Knee
Keywords: knee osteoarthritis; Kinesiotape; Physical performance; Muscle activation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taping group (Experimental): Facilitation taping will be applied to the rectus femoris of patients with knee OA in the taping group.
  Interventions: Other: kinesiology tape
- placebo group (Placebo Comparator): The patients with knee OA in the placebo group will be placed tape on the rectus femoris without any tension.
  Interventions: Other: Placebo tape

INTERVENTIONS:
Other: kinesiology tape — The tape will be fixed without any tension 10 cm below the origin of the rectus femoris muscle. Then 35-50% tension will be applied to the band and descended to the patella. After this point, the Y-shaped band will be terminated to wrap the patella medially and laterally without any tension.
  Arms: taping group
Other: Placebo tape — The tape will attach to the rectus femoris without any tension.
  Arms: placebo group

SUMMARY:
The aim of this study is to determine instant effect of kinesiology taping applied to the rectus femoris on muscle activation, physical performance and proprioception in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
40 patients with knee OA will be included in the study. Intervention group and placebo group will be formed. Facilitation taping will be applied on the rectus femoris of the patients in the taping group. The patients in the placebo group will be placed tape on the rectus femoris without any tension. Muscle activation, physical performance and proprioception will be evaluated before taping and 30 minutes after taping.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45-65 years,
* Patients with independent ambulation,
* Patients with Grade II-III knee osteoarthritis according to the Kellgren and Lawrence Classification,
* Patients not using NSAIDs during the study,
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Patients with previous surgery on the lower extremities
* Patients with neuromuscular disease
* Patients with vestibular pathology
* Patients with diseases of the cardiopulmonary system,
* Patients with communication difficulties,
* Patients who have received physiotherapy or intra-articular injections in the last 6 months or who exercise

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
muscle activation | 5 minutes
  The muscular activation of the Rectus Femoris will be measured with the EMG (Euro Track MyoPlus 4) device before and after the taping application. With the patient in the sitting position with the hip and knee flexed to 90 degrees, active electrodes will be placed on the motor point of the muscle, three measurements will be made, and the highest MVIC value will be recorded.

SECONDARY OUTCOMES:
timed up and go test | 5 minutes
  Individuals will be asked to get up while sitting on the chair, walk three meters, return from the marked point at the end of three meters, walk towards the chair again and sit on the chair. The time taken for the individual's performances will be recorded in seconds.
5 times sit-to-stand test | 1 minutes
  Patients will be asked to stand up and sit down fully upright from the chair with armrests as quickly as possible five times, and the elapsed time will be recorded.
proprioception | 5 minutes
  Participants will sit on a chair with 90° knee flexion. The lower extremities of the participants will be passively and randomly moved from 90° knee flexion to each of the 15°, 30° and 45° angles. After holding the lower extremity at each target angle for 10 seconds, return to the starting position. After waiting 10 seconds in the starting position, the participants will bring their knees to the target angle on their own and stop. Accordingly, the absolute value of the participant's deviation from the target angle will be measured three times for each target angle with the help of a goniometer and the average value will be calculated.
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) | 5 minutes
  It consists of three parts and 24 questions in which pain, stiffness and physical function are questioned. The maximum scores that can be obtained from the index are 20 for the pain subgroup, 8 for stiffness, and 68 for physical function. High scores indicate increased pain and stiffness and impaired physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin ATAŞ, Principal Investigator — Kırıkkale University
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuzun EH, Eker L, Aytar A, Daskapan A, Bayramoglu M. Acceptability, reliability, validity and responsiveness of the Turkish version of WOMAC osteoarthritis index. Osteoarthritis Cartilage. 2005 Jan;13(1):28-33. doi: 10.1016/j.joca.2004.10.010. PMID 15639634
- [Background] Ye W, Jia C, Jiang J, Liang Q, He C. Effectiveness of Elastic Taping in Patients With Knee Osteoarthritis: A Systematic Review and Meta-Analysis. Am J Phys Med Rehabil. 2020 Jun;99(6):495-503. doi: 10.1097/PHM.0000000000001361. PMID 31851010